CLINICAL TRIAL: NCT02184897
Title: Pharmacokinetic and Pharmacodynamic Study of Lenograstim for Hematopoietic Stem Cell Mobilization in Patients With Multiple Myeloma
Brief Title: Pharmacokinetic and Pharmacodynamic Study of Lenograstim for Hematopoietic Stem Cell Mobilization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Cheolwon Suh, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AMC_MM01
Record Dates: First submitted 2014-06-22; First posted 2014-07-09 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AM group (Active Comparator): Lenograstim is administered at 8 am and apheresis is started at 10 am on D4.
  Interventions: Drug: lenograstim 10 microgram/kg/day
- PM group (Experimental): Lenograstim is administered at 6 pm and apheresis is started at 8 am on D5
  Interventions: Drug: lenograstim 10 microgram/kg/day

INTERVENTIONS:
Drug: lenograstim 10 microgram/kg/day

SUMMARY:
Twenty four patients with multiple myeloma will be randomized to either AM group (administration of lenograstim at 8 am) or PM group (administration of lenograstim at 6 am ). Apheresis of hematopoietic stem cell will start at 10 am on D5 in AM group and at 8 am on D4 in PM group, respectively. Pharmacokinetic data of lenograstim will be correlated with pharmacodynamic data of CD34+ cell count, absolute neutrophil cell count and hematopoeitic progenitor cell count. In addition, the yield of stem cell collection between two arms will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* age: above 17 years, below 65 years old
* informed consent
* ECOG 0-1
* autologous stem cell transplant candidate among patients with multiple myeloma

Exclusion Criteria:

* prior history of hematopoetic stem cell transplantation
* history of failure to mobilize hematopoietic stem cells
* history of G-CSF administration within 2 weeks before enrollment to this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-08 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
pharmacokinetic data of lenograstim | on day 1 of apheresis
  AUC0-24hr, Cmax, Cmin, Tmax, T1/2 of lenograstim

SECONDARY OUTCOMES:
pharmacodynamic data: CD34+ cell count by flow cytometry | on day 1 of apheresis
pharmacodynamic data: absolute neutrophil count | on day 1 of apheresis
pharmacodynamic data: hematopoietic progenitor cells (HPC) | on day 1 of apheresis

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Asan Medical Center, University of Ulsan College of Medicine, Seoul
  - Asan Medical Center, Seoul